CLINICAL TRIAL: NCT00549042
Title: A Phase III, Variable-Dose Titration Followed by a Randomized Double-Blind Study of Controlled-Release OROS® Hydromorphone HCl (NMED-1077) Compared to Placebo in Patients With Chronic Low Back Pain
Brief Title: Study to Test the Effectiveness of Controlled-Release OROS® Hydromorphone HCl Compared to Placebo in Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMT 1077-301
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2019-02

CONDITIONS: Chronic Low Back Pain
Keywords: Back Pain; Chronic Low Back Pain; Chronic Back Pain; Pain; Chronic Pain
MeSH Terms: conditions — Back Pain; Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- OROS hydromorphone (Experimental): OROS hydromorphone tablets administered orally once daily in total daily doses of 12, 16, 24, 32, 40, 48, or 64 mg
  Interventions: Drug: OROS hydromorphone
- placebo (Placebo Comparator): Matching placebo tablets orally once daily (number and dosage of tablets to match the number and dosage of the stable dose of OROS hydromorphone obtained in the Conversion and Titration phase).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OROS hydromorphone — hydromorphone 12, 16, 24, 32, 40, 48, or 64 mg tablets
  Arms: OROS hydromorphone
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This study will test an experimental drug called OROS® hydromorphone hydrochloride (HCl) (NMED-1077), a once daily opioid analgesic that can relieve pain. A large number of clinical studies have been conducted to test this drug. OROS hydromorphone HCl is currently approved in both the US and Europe to treat chronic pain.

The purpose of this study is to compare OROS hydromorphone to placebo to see if it is safe and efficacious.

ELIGIBILITY:
Inclusion Criteria

1. Patients must have been provided with written consent to participate in the study prior to any study procedures, and must understand that they are free to withdraw from the study at any time.
2. Patients who can speak, read, write, and understand English, and must be able to read and understand the consent form, complete study-related procedures, and communicate with the study staff.
3. Male and female patients aged 18-75 years, inclusive.
4. Documented diagnosis of moderate to severe chronic low back pain that must have been present
5. Patients who are classified as non-neuropathic (Class 1 and 2) or neuropathic (Class 3, 4, 5 and 6) of lower back pain based on the Quebec Task Force Classification of Spinal Disorders will be enrolled for this study.
6. Patients who require daily scheduled opioid analgesics for low back pain for at least 2 months prior to the screening visit.
7. Patients with a daily opioid requirement of ≥ 60 mg oral morphine equivalent (≥ 12 mg hydromorphone), but ≤ 320 mg morphine (≤ 64 mg hydromorphone) per day within the 2 months prior to the screening visit.
8. Patients who, in the Investigator's opinion, are on a stable dose (≥ 2 weeks) of all prior analgesics (both opioid and non-opioid) prior to the screening visit.
9. Female subjects of childbearing potential including those who have had a tubal ligation surgery but excluding those who have not experienced a menstrual period for a minimum of 2 years, must have a negative serum pregnancy test at screening visit, and must consent to utilize a medically acceptable method of contraception throughout the entire study period including the washout period and for 1 week after the study is completed.

Exclusion Criteria

1. Patients with an active diagnosis of fibromyalgia, complex regional pain syndrome (including reflex sympathetic dystrophy or causalgia), acute spinal cord compression, severe or progressive lower extremity weakness or numbness, bowel or bladder dysfunction as a result of cauda equina compression, diabetic amyotrophy, meningitis, diskitis, back pain because of secondary infection or tumor, or pain caused by a confirmed or suspected neoplasm.
2. Patients who have undergone a surgical procedure for back pain within 6 months prior to the screening visit.
3. Patients who have had nerve or plexus block, including epidural steroid injections or facet blocks, within 1 month prior to the screening visit.
4. Patients with any other chronic pain condition that, in the investigator's opinion, would interfere with the assessment of low back pain (e.g., osteoarthritis, rheumatoid arthritis, postherpetic neuralgia, pain associated with diabetic neuropathy, migraine headaches requiring opioid therapy).
5. Patients who are involved in an active workman's compensation or insurance claim or disability claim or litigation related to back pain.
6. Patients who have by history used any illicit drugs of abuse, abused opioids or exhibited drug seeking behavior within 5 years prior to the screening visit.
7. Patients who have abused prescription medication or alcohol within 5 years prior to the screening visit.
8. Patients with a positive alcohol or drugs of abuse test
9. Women who are pregnant (as indicated by a positive result in a serum pregnancy test administered at screening visit), or breast feeding, or planning to breast feed within 30 days prior to the screening visit.
10. Patients who have demonstrated allergic reactions or hypersensitivity to opioids.
11. Patients who have had no bowel movement within three days, or bowel obstruction within 60 days, prior to the screening visit.
12. Patients with pre-existing severe narrowing of the gastrointestinal tract secondary to:

    prior gastrointestinal surgery (e.g., vagotomy, antrectomy, pyloroplasty, gastroplasty, gastrojejunostomy) or gastrointestinal disease resulting in impaired gastrointestinal function (e.g., paralytic ileus, gastroparesis, inflammatory bowel disease, "short gut" syndrome due to adhesions or decreased transit time, past history of peritonitis, cystic fibrosis, chronic intestinal pseudoobstruction, or Meckel diverticulum)
13. Patients who have a major psychiatric condition (e.g., schizophrenia, major depression) or who have clinically significant anxiety or depression as defined by a Hospital Anxiety and Depression Scale(HADS) score greater than 10.
14. Patients who have received monoamine oxidase (MAO) inhibitors within 14 days prior to the screening visit.
15. Patients with clinically significant abnormal laboratory results in clinical chemistry, hematology or urinalysis including serum glutamic-oxaloacetic transaminase/aspartate aminotransferase (AST) or serum glutamic-pyruvic transaminase/alanine aminotransferase (ALT) ≥ 3.0 times the upper limit of the reference range or a serum creatinine ≥ 2.0 mg/dL at screening.
16. Patients with a serious or unstable intercurrent illness.
17. Patients with a history of uncontrolled seizure disorder.
18. Patients with increased intracranial pressure, mental clouding of unknown etiology, coma, or hypotension.
19. Patients who have severe asthma, severe chronic obstructive pulmonary disease, or any other disorder that predisposes the patient to carbon dioxide retention or respiratory depression.
20. Patients who have taken any investigational drug within 30 days prior to the screening visit or are currently enrolled in another investigational drug study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

REFERENCES:
- [Derived] Nalamachu S, Hale M, Khan A. Hydromorphone extended release for neuropathic and non-neuropathic/nociceptive chronic low back pain: a post hoc analysis of data from a randomized, multicenter, double-blind, placebo-controlled clinical trial. J Opioid Manag. 2014 Sep-Oct;10(5):311-22. doi: 10.5055/jom.2014.0221. PMID 25350473
- [Derived] Hale M, Khan A, Kutch M, Li S. Once-daily OROS hydromorphone ER compared with placebo in opioid-tolerant patients with chronic low back pain. Curr Med Res Opin. 2010 Jun;26(6):1505-18. doi: 10.1185/03007995.2010.484723. PMID 20429852

RESULTS

PARTICIPANT FLOW:
Period: Conversion and Titration Phase
Arm/Group | OROS Hydromorphone | Placebo
Started | 459 | 0 (Per the study design, no patients received placebo during this phase.)
Completed | 268 | 0 (Per the study design, no patients received placebo during this phase.)
Not Completed | 191 | 0
Period: Double-blind Phase
Arm/Group | OROS Hydromorphone | Placebo
Started (Patients who completed titration and conversion were allowed in the double-blind phase.) | 134 | 134
Completed | 66 | 44
Not Completed | 68 | 90

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OROS Hydromorphone | Placebo | Total
Number analyzed (Participants) | 134 | 134 | 268
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 123 | 252
  >=65 years | 5 | 11 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.51) | 49.5 (10.55) | 48.6 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 73 | 134
  Male | 73 | 61 | 134
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 134 | 134 | 268

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Mean Pain Intensity
Description: Participants rate their pain intensity on a numeric rating scale (NRS), where 0=no pain and 10=worst possible pain, in a daily diary. At Week 12 (or final visit), all measurements during the preceding week are averaged, and the mean change from the mean score at baseline is calculated.
Time Frame: Baseline, Week 12 (or final visit)
Population: Intent-to-treat population (ITT). One patient (randomized to receive OROS hydromorphone) did not report taking any study medication, and another (randomized to receive placebo) did not have Baseline values for the primary efficacy variable; both were excluded from the ITT population. Therefore, the ITT population had 266 patients.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | OROS Hydromorphone | Placebo
Number analyzed (Participants) | 133 | 133
score on a scale | 0.6 [-5 to 5] | 1.7 [-3 to 7]

2. Other Pre Specified Outcome: Change From Baseline in Mean Pain Intensity Scores Through the Entire 12-week Treatment Phase
Description: Participants rate their pain on the pain intensity NRS in a daily diary. At each scheduled visit all measurements during the preceding week are collected, and a mean score for each arm is calculated for each visit. Mean scores at baseline and each subsequent visit are plotted on a graph for the entire 12-week treatment period, and an area under the curve calculation is used to determine the mean change from baseline for each arm through the entire 12-week treatment phase.
Time Frame: Baseline through Week 12
Population: Results are not presented for Other, prespecified outcome measures
Arm/Group | OROS Hydromorphone | Placebo
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Change From Baseline in Mean Patient Global Assessment (PGA) Scores
Description: Change from Baseline in mean PGA scores collected at each visit (at Baseline, Days 1, 4, 8, 11, and Weeks 2, 3, 4, 6, 8, 10, and 12) using the scale: 1=Excellent, 2=Very Good, 3=Good, 4=Fair, and 5=Poor. The worst possible score is 5.0.
Time Frame: Baseline through Week 12
Population: Results are not presented for Other, prespecified outcome measures
Arm/Group | OROS Hydromorphone | Placebo
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Change From Baseline in Mean Scores on the Roland-Morris Disability Questionnaire
Description: Change from baseline in the Roland-Morris Disability Questionnaire (RDQ) score was analyzed for each visit at which the RDQ was administered (Days 1, 8, and Weeks 2, 3, 4, 6, 8, 10, and 12). This is a 24-item inventory with scores ranging from 0 (highest ability) to 24 (lowest ability). Higher scores mean more disability.
Time Frame: Baseline through Week 12
Population: Results are not presented for Other, prespecified outcome measures
Arm/Group | OROS Hydromorphone | Placebo
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Change From Baseline in Mean Pain Intensity Scores Collected at Scheduled Visits to the Clinic
Description: Participants rate their pain on the pain intensity NRS at each scheduled visit (Baseline, Days 1, 4, 8, 11, and Weeks 2, 3, 4, 6, 8, 10, and 12), and a mean score is calculated.
Time Frame: Baseline through Week 12
Population: Results are not presented for Other, prespecified outcome measures
Arm/Group | OROS Hydromorphone | Placebo
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Time to Treatment Failure
Description: Time to treatment failure is the median number of days from baseline until the earliest day on which the patient's data indicated treatment failure.
Time Frame: within 12 weeks
Population: Results are not presented for Other, prespecified outcome measures
Arm/Group | OROS Hydromorphone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The safety population includes all patients who were enrolled and who took at least one dose of study drug (N=447). Adverse event displays include data from the safety population. The number of subjects who entered the Conversion and Titration phase was 459.
Groups:
- Conversion and Titration Phase: OROS hydromorphone 12, 16, 24, 32, 40, 48, or 64 m
Arm/Group | Conversion and Titration Phase | OROS Hydromorphone | Placebo
Serious Adverse Events (participants affected / at risk) | 5/447 | 6/134 | 4/134
Other Adverse Events (participants affected / at risk) | 247/447 | 64/134 | 73/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conversion and Titration Phase (N=447) | OROS Hydromorphone (N=134) | Placebo (N=134)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosi (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Possible kidney stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conversion and Titration Phase (N=447) | OROS Hydromorphone (N=134) | Placebo (N=134)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 3
Toothache (Gastrointestinal disorders) | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 69 | 10 | 5
Diarrhoea (Gastrointestinal disorders) | 13 | 5 | 9
Dry mouth (Gastrointestinal disorders) | 13 | 0 | 0
Nausea (Gastrointestinal disorders) | 53 | 12 | 10
Vomiting (Gastrointestinal disorders) | 29 | 8 | 6
Chills (General disorders) | 0 | 2 | 3
Pain (General disorders) | 0 | 1 | 3
Drug withdrawal syndrome (General disorders) | 22 | 13 | 16
Fatigue (General disorders) | 16 | 1 | 4
Oedema peripheral (General disorders) | 13 | 3 | 1
Influenza (Infections and infestations) | 0 | 4 | 2
Sinusitis (Infections and infestations) | 0 | 6 | 1
URT infection (Infections and infestations) | 0 | 4 | 3
Urinary tract infection (Infections and infestations) | 0 | 4 | 2
Weight decreased (Investigations) | 0 | 4 | 3
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 8 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 6 | 8
Tremor (Nervous system disorders) | 0 | 1 | 3
Dizziness (Nervous system disorders) | 17 | 3 | 2
Headache (Nervous system disorders) | 35 | 7 | 10
Somnolence (Nervous system disorders) | 39 | 0 | 0
Anxiety (Psychiatric disorders) | 9 | 0 | 4
Insomnia (Psychiatric disorders) | 13 | 3 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 13 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No